CLINICAL TRIAL: NCT03800628
Title: Perception of Quality of Life and Resource Availability After Surviving Critical Illness
Brief Title: Resource Availability Following Critical Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Walden University (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Michelle McMoon, Principle Investigator, Walden University
Other Study IDs: 09-06-2018-0576535
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Quality of Life
Keywords: survivor; QOL; resources

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: qualitative study — semi-structured interviews

SUMMARY:
The purpose of this qualitative study is to explore the vital issues in recovery of QOL from the perspective of survivors of critical illness and understand these patients' views on rehabilitative services in the United States (U.S.). The theoretical framework for this study is Max Weber's Rational Choice Theory (RCT). The research questions will focus on understanding post-ICU QOL and the patients' experience with rehabilitative services following critical illness. A phenomenological study design is being employed, using semi-structured individual interviews with critical illness survivors. Data from the interviews will be coded for thematic analysis. The implications for social change include defining the meaning of QOL for an ICU survivor and improving healthcare policies for the therapies necessary to return survivors to a life worth living.

DETAILED DESCRIPTION:
The purpose of this qualitative study is to understand the patient perception of QOL after surviving critical illness and how survivors can help illuminate gaps in current health policies to provide better recovery resources for this growing population.

The central research questions are:

RQ1: What are the issues important to preserve quality of life from the perspective of critical illness survivors? RQ2: How do survivors of critical illness describe rehabilitative services after discharge?

ELIGIBILITY:
Inclusion Criteria:

* critical illness survivors within 18 months of ICU discharge
* minimum 48 hours of mechanical ventilation
* ability to read and understand English
* over the age of 18

Exclusion Criteria:

* emotional or psychological inability to participate in a 30-min interview
* not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critical illness survivors
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
RQ1: What are the issues important to preserve quality of life from the perspective of critical illness survivors? | 6 months
  semi-structured, open-ended qualitative interview

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided